CLINICAL TRIAL: NCT00122265
Title: Exploring Genomic, Proteomic and Dosimetric Determinants of Late Toxicity After Three Dimensional Conformal RT for Prostate Cancer
Brief Title: Exploring Genomic, Proteomic and Dosimetric Determinants of Late Toxicity After Three Dimensional Conformal Radiotherapy (RT) for Prostate Cancer
Status: Terminated | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: GU-6-0035/ethics 17075
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radiotherapy; radiation toxicity; single nucleotide polymorphism
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prostate cancer is the most common malignancy in males, and radiotherapy is a commonly chosen treatment option for patients with localized disease. Technical innovations such as three-dimensional conformal radiotherapy (3D CRT) and intensity-modulated radiotherapy permit radiation dose escalation and possibly better disease outcomes, but escalated doses may be accompanied by long-term complications. This study will examine, for the first time, the independent contribution of a patient's own genetic makeup to the development of post-radiation complications, permitting the future development of predictive tests to avoid radiation injury. To do this, the investigators will examine gene markers and blood proteins in a series of approximately 100 prostate cancer survivors who have received three-dimensional conformal radiotherapy between 1996 and 2000 at the Cross Cancer Institute.

DETAILED DESCRIPTION:
OBJECTIVES: Major innovations in radiotherapy (RT) delivery (3D conformal RT, intensity modulated RT) now permit RT dose escalation to be tested as a means of improving control of localized prostate cancer. With delivery innovations, severe toxicity occurs rarely, but significant bladder and rectal toxicity is common. The investigators have studied a cohort of 98 patients who received dose-escalated 3D-CRT and have obtained evidence of dosimetric factors underlying rectal toxicity. They posit that the late radiation toxicity disease state has significant genetic determinants. These determinants are neither understood nor accounted for in selection of treatment, and the investigators propose to study the above well-characterized cohort, who are clinically well from a disease control perspective, given that comprehensive dosimetric and outcome information is available on all.

HYPOTHESIS: Comprehensive analysis of the genomic, proteomic, and dosimetric characteristics of patients with prostate cancer will provide a novel understanding of the genetic predisposition of cellular and tissue responses to irradiation which result in the clinical occurrence of significant chronic rectal and bladder injury after 3D-CRT.

APPROACH: For a thorough understanding of the molecular processes underlying tissue responses to radiation damage, the investigators propose a genomic analysis. Their working hypothesis is that rectal and bladder toxicity will be correlated to patient genetics as measured by single nucleotide polymorphisms (SNPs) in a select group of genes. The criteria for selecting SNPs will be based on evidence for the various genes implicated or demonstrated in DNA repair pathways and radiation-induced tissue damage. In addition, since radiation injury can be considered a phenotypic tissue response to RT in genetically predisposed individuals, the investigators will examine the protein profile "signature" in sera from patients who have suffered significant toxicity. Analysis of these data will be unique in that the investigators will use both statistically based bioinformatics approaches, and biophysical modeling. This proposal represents the most comprehensive exploration to date of the concept of a molecular "signature" of normal tissue radiation injury of which the applicants are aware.

SPECIFIC AIM 1:

* To create a database of SNPs among long-term prostate cancer survivors who have been treated with 3D-CRT, and for whom detailed toxicity, quality of life and dosimetric information are available;
* To assess the feasibility of using bioinformatics approaches with this database to examine the possibility that specific SNPs, in the context of known dosimetric factors, can predict occurrence of late rectal or bladder toxicity;
* To perform a proteomic analysis of serum samples from a cohort of 25 patients experiencing higher levels of ongoing late toxicity and 50 patients with no ongoing late toxicity.

SPECIFIC AIM 2:

* To utilize biophysical approaches to modelling clinical complication data, using the concept of generalized mean biological effective dose (GMBED) and the critical volume model.

SUMMARY: This proposal will be the first comprehensive retrospective analysis of genomic, proteomic and dosimetric determinants of late radiation injury in prostate cancer. The investigators have assembled a broad array of expertise from the CCI PolyomX program (the only high throughput SNP facility in western Canada), the NCI/FDA Clinical Proteomics Program at Bethesda, MD, and the unique biophysical modeling capability of CBIAR researchers to reach these goals.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with 3D CRT for which follow-up toxicity evaluation was done

Exclusion Criteria:

* Follow-up less than 18 months

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2003-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Parliament, MD, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada